CLINICAL TRIAL: NCT03299985
Title: Effects of Diaphragmatic Myofascial Release in Gastroesophageal Reflux Disease
Brief Title: Diaphragmatic Myofascial Release in Gastroesophageal Reflux Disease
Acronym: GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of medicine department, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JParraga
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux Disease; Myofascial release; Diaphragm
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: double blinded randomized clinical trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic myofascial release (Experimental): Subjects in this arm will receive different myofascial release techniques aimed to normalize the myofascial tension of the diaphragmatic muscle
  Interventions: Other: Diaphragmatic myofascial release
- Sham myofascial release (Sham Comparator): Subjects in this arm will receive the same manual techniques of the diaphragmatic myofascial release group, but without the myofascial stimulus
  Interventions: Other: Sham myofascial release

INTERVENTIONS:
Other: Diaphragmatic myofascial release — Subjects in this arm will receive different myofascial release techniques aimed to normalize the myofascial tension of the diaphragmatic muscle
  Arms: Diaphragmatic myofascial release
Other: Sham myofascial release — Subjects in this arm will receive the same manual techniques of the diaphragmatic myofascial release group, but without the myofascial stimulus
  Arms: Sham myofascial release

SUMMARY:
This study is a double blinded randomized clinical trial with two arms which aims to study the effects of diaphragmatic myofascial release in patients with gastroesophageal reflux disease (GERD).

GERD has become in the last decades a common disease at the occidental world affecting between 10 to 15% of this population. That implies a high socio-health cost and the decline of the quality of life of those patients.

The diaphragm muscle surrounds the lower esophageal sphincter, and helps to prevent gastroesophageal reflux. If one or both structures become incompetent, it may appear GERD. Until the moment, the treatment for GERD begins by lifestyle modification, and if it fails, the treatment becomes medical and, in selected cases, surgical.

It exists some studies that have demonstrate that diaphragmatic breathing training can have a positive effect in GERD and the need of drug usage. But until the moment, the effects of a myofascial release of the diaphragm haven't been explored on these patients.

Thirty patients with GERD referred from different hospitals of Valencia will be randomized into two groups:

* Intervention with myofascial release for the diaphragm
* Sham treatment group which is going to receive the same number of session treatments with the same manual techniques, but without the myofascial stimulus The protocol that will be applied consists of 4 identical sessions of myofascial release techniques aimed to normalize the myofascial tension of the diaphragmatic muscle. These sessions will be distributed in two weeks.

The study focuses on the analysis of the following variables:

* Frequency and intensity of the symptoms of GERD: Reflux Disease Questionnaire (RDQ)
* Specific quality of life for gastrointestinal disease: Gastrointestinal Quality of life Index (GIQLI)
* Drug usage: weekly milligrams usage of proton pomp inhibitors (PPI) The results of these pre-intervention and post-intervention variables will be compared between the two groups at baseline (first session), at week 3 and at week 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnostic of GERD

Exclusion Criteria:

* hiatal hernia >2 cm
* previous operation at the LES
* actual erosive esophagitis
* Congenital or acquired immune disorders.
* Allergic status of any kind.
* Systemic diseases (rheumatic, infectious conditions, febrile state, vascular alterations, endocrine including diabetes, metabolic and neoplastic).
* Leukemia.
* Severe psychiatric disorders.
* Neuromuscular or neurological injuries.
* Aneurysms.
* Abdominal or spine surgery.
* Vertebral fractures.
* Osteoporosis (advanced stage).
* Acute lesions of soft tissues or in an inflammatory state.
* Open wounds.
* Pregnancy.
* Intrauterine device.
* Patients with corticosteroid therapy.
* Hemophilia or treatment with anticoagulant therapy.
* Hypersensitivity of the skin or dermatological diseases in the trunk that impossibilities the application of the techniques.
* Rejection of manual contact.
* Non-Spanish speaking patients.
* Patients who have previously received some treatment of myofascial release.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
GERD symptoms | 6 weeks
  Frequency and intensity of GERD symptoms measured by the Reflux Disease questionnaire (RDQ)

SECONDARY OUTCOMES:
Specific quality of life for gastrointestinal disease | 6 weeks
  Gastrointestinal Quality of life Index (GIQLI)
Drug Usage | 6 weeks
  Weekly milligrams usage of proton pomp inhibitors (PPI)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Quintana JM, Cabriada J, Lopez de Tejada I, Varona M, Oribe V, Barrios B, Perdigo L, Bilbao A. Translation and validation of the gastrointestinal Quality of Life Index (GIQLI). Rev Esp Enferm Dig. 2001 Nov;93(11):693-706. English, Spanish. PMID 11995369
- [Background] Shaw M, Dent J, Beebe T, Junghard O, Wiklund I, Lind T, Johnsson F. The Reflux Disease Questionnaire: a measure for assessment of treatment response in clinical trials. Health Qual Life Outcomes. 2008 Apr 30;6:31. doi: 10.1186/1477-7525-6-31. PMID 18447946
- [Background] Nuevo J, Tafalla M, Zapardiel J. [Validation of the Reflux Disease Questionnaire (RDQ) and Gastrointestinal Impact Scale (GIS) in patients with gastroesophageal reflux disease in the Spanish population]. Gastroenterol Hepatol. 2009 Apr;32(4):264-73. doi: 10.1016/j.gastrohep.2008.12.004. Epub 2009 Apr 16. Spanish. PMID 19371971
- [Result] da Silva RC, de Sa CC, Pascual-Vaca AO, de Souza Fontes LH, Herbella Fernandes FA, Dib RA, Blanco CR, Queiroz RA, Navarro-Rodriguez T. Increase of lower esophageal sphincter pressure after osteopathic intervention on the diaphragm in patients with gastroesophageal reflux. Dis Esophagus. 2013 Jul;26(5):451-6. doi: 10.1111/j.1442-2050.2012.01372.x. Epub 2012 Jun 7. PMID 22676647
- [Result] Eherer AJ, Netolitzky F, Hogenauer C, Puschnig G, Hinterleitner TA, Scheidl S, Kraxner W, Krejs GJ, Hoffmann KM. Positive effect of abdominal breathing exercise on gastroesophageal reflux disease: a randomized, controlled study. Am J Gastroenterol. 2012 Mar;107(3):372-8. doi: 10.1038/ajg.2011.420. Epub 2011 Dec 6. PMID 22146488
- [Result] Arguisuelas MD, Lison JF, Sanchez-Zuriaga D, Martinez-Hurtado I, Domenech-Fernandez J. Effects of Myofascial Release in Nonspecific Chronic Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 May 1;42(9):627-634. doi: 10.1097/BRS.0000000000001897. PMID 28441294